CLINICAL TRIAL: NCT00997815
Title: The Randomized Double-blind Placebo-controlled Trial of Intralesional Botulinum Toxin A Injection for Recalcitrant Alopecia Totalis and Alopecia Universalis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Rattapon Thuangtong, Assistant professor, Siriraj Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: SirirajH
Record Dates: First submitted 2009-10-18; First posted 2009-10-19 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Recalcitrant Alopecia Totalis; Recalcitrant Alopecia Universalis
Keywords: Recalcitrant; Alopecia totalis; Alopecia universalis; Botulinum toxin A
MeSH Terms: conditions — Alopecia universalis | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin A (Experimental): The area of alopecia is splited into experimental and control sides by blocked randomization. Experimental sides injected with botulinum toxin A at 2 units per 0.1 ml of dilution with normal saline entire all area.
  Interventions: Drug: Botulinum toxin A
- Placebo (Placebo Comparator): Using normal saline
  Interventions: Drug: Normal saline injection

INTERVENTIONS:
Drug: Botulinum toxin A — Concentration at 2 units per 0.1 of normal saline dilution
  Other Names: Botox
  Arms: Botulinum toxin A
Drug: Normal saline injection — Using normal saline 2.5 ml injected in control side
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine the efficacy of intralesional botulinum toxin type A injection for recalcitrant alopecia totalis and alopecia universalis.

Treatments of recalcitrant alopecia totalis and universalis remains an challenge issue for medical practice.The application of diphenylcyclopropenone (DPCP) is still being an standard treatment for the condition, however, there are at least thirty percentage of patients recalcitrant to this treatment.

The complete etiology of this disease has yet to be clear.Nevertheless,recent studies have demonstrated the hypothesis of neurotransmitter involvements.

There is numerous evidence in support of an imbalance of transmitters, including substance P and Calcitonin gene-related peptide.

Botulinum toxin A injection has been used to treat a neuralgiform headache and diffused alopecia areata. Both headache and hair loss have been made much in improvement. This data may support the neurotransmitter imbalance theory.

The investigators have been informed about possible effects to the alopecia condition, therefore, this study is conducted to assess the efficacy of botulinum toxin A as the novel treatment for recalcitrant alopecia totalis and alopecia universalis.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be over 18 years old
2. All patients are diagnosed with alopecia totalis or alopecia universalis
3. The alopecia condition was not responded to any treatments

Exclusion Criteria:

1. Having an active inflammation on scalp area
2. Allergic to botulinum toxin A of human albumin
3. Has been diagnosed with neuromuscular disorders
4. Taking any medication that may interfere with botulinum toxin A action
5. Receiving any treatment for alopecia condition within 4 weeks
6. Pregnant , breastfeeding, plan to pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the percentage of terminal hair regrowth in recalcitrant alopecia totalis and alopecia universalis after intralesional botulinum toxin A injection | 4 months

SECONDARY OUTCOMES:
To evaluate any possible side effects of intralesional botulinum toxin A injection for alopecia totalis and alopecia universalis | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Rattapon Thoungtong, MD, Study Chair — Department of Dermatology, Faculty of medicine Siriraj Hospital, Mahidol University; Supenya Varothai, MD, Study Director — Department of Dermatology, Faculty of Medicine Siriraj Hospital, Mahidol University; Rasthawathana Desomchoke, MD, Principal Investigator — Department of Dermatology, Faculty of Medicine Siriraj Hospital, Mahidol University; Suthasinee Pattaravadee, B.Sc, Principal Investigator — Department of Dermatology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Department of dermatology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand